CLINICAL TRIAL: NCT00703313
Title: Ocular Availability in Human Tears After Topical Administration of 1.5% Levofloxacin Compared to Active Comparators
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Brian Schwam, MD/Medical Director, VISTAKON Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VPH0108
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Study drug concentration in human tears

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2 (Active Comparator): described in intervention
  Interventions: Drug: 0.5% moxifloxacin hydrochloride ophthalmic solution
- 3 (Active Comparator): described in intervention
  Interventions: Drug: 0.3% gatifloxacin ophthalmic solution
- 1 (Active Comparator): described in intervention
  Interventions: Drug: 1.5% levofloxacin ophthalmic solution

INTERVENTIONS:
Drug: 1.5% levofloxacin ophthalmic solution — 1 drop instilled at each visit
  Arms: 1
Drug: 0.5% moxifloxacin hydrochloride ophthalmic solution — 1 drop instilled at each visit
  Arms: 2
Drug: 0.3% gatifloxacin ophthalmic solution — 1 drop instilled at each visit
  Arms: 3

SUMMARY:
The primary objective of this study is to compare the concentration in human tears of levofloxacin and the active comparators at 15 minutes, 2,6, 12, and 24 hours after instillation of a single drop of medication.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent and HIPAA indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Be willing and able to follow all instructions and attend all study visits
* If female and of childbearing potential, not be pregnant, nursing or planning a pregnancy and agree to submit to a pregnancy test. The result of the test must be negative and female subjects of childbearing potential must also agree to use an acceptable method of contraception for the duration of the study (acceptable method of contraception includes oral, implantable, transdermal, or injectible contraceptives, spermicide with barrier, IUD, or surgical sterilization of partner)

Exclusion Criteria:

* Have a known allergy and/or sensitivity to the test article(s) or its components or any therapies associated with the study
* Have active signs or symptoms of any clinically significant ocular disorder (other than refractive disorders)
* Have a history of dry eye syndrome
* Use disallowed medications (systemic or topical) (i.e. any fluoroquinolone anti-infective agents or any topical ophthalmic products) during the appropriate pre-study washout period and during the study.
* Be a contact lens wearer who is unwilling to forego contact lens wear within 3 days prior to the start of the study and for the duration of the study
* Have had any ocular surgical intervention 12 months prior to the study or anticipate having ocular surgery during the study
* Be pregnant or nursing women; or women who have a positive urine pregnancy test at screening or women of childbearing potential who refuse to use an adequate hormonal or mechanical means of birth control
* Be concurrently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of entry into this study
* Employees of the investigator or study center, with direct involvement in th proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Concentration of levofloxacin, moxifloxacin or gatifloxacin in tears | 15 minutes, 2, 6, 12 and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Vistakon, Jacksonville, Florida, United States